CLINICAL TRIAL: NCT05950464
Title: A Phase 1B Study of Combination ATR (M1774) and BET Inhibition (ZEN003694) to Exploit ARID1A Loss in Recurrent Ovarian and Endometrial Cancer
Brief Title: Testing Different Amounts of the Combination of Drugs M1774 and ZEN-3694 for the Treatment of Recurrent Ovarian and Endometrial Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2023-03408; NCI-2023-03408 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY031 (Other: NRG Oncology); NRG-GY031 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2023-07-15; First posted 2023-07-18 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Endometrial Carcinoma; Recurrent Endometrial Clear Cell Adenocarcinoma; Recurrent Endometrial Endometrioid Adenocarcinoma; Recurrent Endometrial Low Grade Endometrioid Adenocarcinoma; Recurrent Ovarian Clear Cell Adenocarcinoma; Recurrent Ovarian Endometrioid Adenocarcinoma; Recurrent Ovarian High Grade Serous Adenocarcinoma; Recurrent Ovarian Low Grade Endometrioid Adenocarcinoma; Recurrent Platinum-Resistant Ovarian Carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Biopsy; Specimen Handling; Magnetic Resonance Spectroscopy; X-Rays; Phantoms, Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (tuvusertib, BET bromodomain inhibitor ZEN-3694) (Experimental): Patients receive tuvusertib and BET bromodomain inhibitor ZEN-3694 PO on study. Patients in the dose-escalation phase of the trial also undergo ECG during screening, collection of blood samples on study, and x-ray, CT, or MRI throughout the trial. Patients in the dose-expansion phase of the trial also undergo ECG during screening, biopsies during screening and on study, and x-ray, CT, or MRI, and collection of blood samples throughout the trial.
  Interventions: Drug: BET Bromodomain Inhibitor ZEN-3694; Procedure: Biopsy Procedure; Procedure: Biospecimen Collection; Procedure: Computed Tomography; Procedure: Electrocardiography; Procedure: Magnetic Resonance Imaging; Drug: Tuvusertib; Procedure: X-Ray Imaging

INTERVENTIONS:
Drug: BET Bromodomain Inhibitor ZEN-3694 — Given PO
  Other Names: BETi ZEN-3694; ZEN 3694; ZEN-3694; ZEN003694
Procedure: Biopsy Procedure — Undergo biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Electrocardiography — Undergo ECG
  Other Names: ECG; EKG
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI
Drug: Tuvusertib — Given PO
  Other Names: ATR Kinase Inhibitor M1774; M 1774; M-1774; M1774
Procedure: X-Ray Imaging — Undergo x-ray
  Other Names: Conventional X-Ray; Diagnostic Radiology; Medical Imaging, X-Ray; Plain film radiographs; Radiographic Imaging; Radiographic imaging procedure (procedure); Radiography; RG; Static X-Ray; X-Ray

SUMMARY:
This phase Ib trial tests the safety, side effects, and best dose of M1774 when given with ZEN-3694 in treating patients with ovarian and endometrial cancer that has come back (recurrent). M1774 and ZEN-3694 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. M1774 and ZEN-3694 combined together has demonstrated to be better than either drug alone in killing ovarian tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) and the dose-limiting toxicities (DLTs) for combination of tuvusertib (ATR inhibitor [M1774]) and BET bromodomain inhibitor ZEN-3694 (BET inhibitor [ZEN003694]) in women with recurrent clear cell, endometrioid, and platinum resistant high grade serous ovarian carcinoma (HGSOC) and clear cell and endometrioid endometrial carcinoma irrespective of ARID1A status (PART I).

II. To determine safety and tolerability in ARID1A pathogenic alteration (ARID1A^MUTATION [MUT]) and ARID1A wildtype (ARID1A^WT) cohorts (ARID1A is an integral biomarker) in an expansion phase (PART II).

III. To determine change in pharmacodynamic biomarker expression of gammaH2AX (for ATR inhibition, integral biomarker) from pre-treatment and on-treatment tumor samples in ARID1A^MUT and ARID1A^WT expansion cohorts by immunohistochemistry (IHC) (PART II).

SECONDARY OBJECTIVES:

I. To evaluate change in pharmacodynamic biomarker expression of cmyc (for BET inhibition, integrated biomarker) from pre-treatment and on-treatment tumor samples in ARID1A^MUT and ARID1A^WT expansion cohorts by Digital Spatial Profiling (DSP) (PART II).

II. To evaluate change in pharmacodynamic biomarker expression of gammaH2AX (for ATR inhibition, integrated biomarker) from pre-treatment and on-treatment tumor samples in ARID1A^MUT and ARID1A^WT expansion cohorts by DSP (PART II).

III. To investigate if ARID1A protein by IHC and DSP correlates with ARID1A pathogenic alteration in pre-treatment tumor biopsy samples (PART II).

IV. To estimate objective response rate (ORR) and progression free survival (PFS) at 6 months in ARID1A pathogenic alteration and wildtype cohorts (PART II).

EXPLORATORY OBJECTIVES:

I. To evaluate the pharmacokinetics of ZEN003694 and its active metabolite, ZEN003791, when the drug is taken alone and in combination with M1774, as well as M1774 pharmacokinetics in the combination (PART I).

II. To assess if ARID1A pathogenic alteration status by Next Generation Sequencing (NGS) correlates with ARID1A protein by IHC utilizing existing archival tissue and evaluate retrospectively (PART I).

III. To evaluate objective response rate (ORR) and progression free survival (PFS) at 6 months and to evaluate if these correlate with ARID1A pathogenic alteration status by Next Generation Sequencing (NGS) and with ARID1A protein by IHC (PART I).

IV. In patients with prior somatic tumor testing by Next Generation Sequencing, will obtain results and correlate molecular profiles (i.e., ARID1A pathogenic alteration, PIK3CA pathogenic alteration, C-myc amplification, ATM pathogenic alteration) with response by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or CA-125 by Gynecological Cancer Intergroup (GCIG) (Rustin et al., 2011) (PART I).

V. To evaluate the pharmacokinetics of ZEN003694 and its active metabolite, ZEN003791, when the drug is taken alone and in combination with M1774, as well as M1774 pharmacokinetics in the combination (PART II).

VI. To assess if there is a greater overall response by RECIST 1.1 and CA-125 by GCIG (Rustin et al. 2011) in ARID1A pathogenic alteration cohort (ARID1A^MUT ) compared to ARID1A wildtype (ARID1A^WT ) cohort (PART II).

VII. To correlate pharmacodynamics and pharmacokinetics in ARID1A^MUT and ARID1A^WT expansion cohorts at the MTD (determine if drug levels affect drug target engagement and expression (e.g., gamma [g]H2AX and MYC)) (PART II).

VIII. To estimate overall survival (OS) in ARID1A pathogenic alteration versus (vs) wildtype cohorts (PART II).

IX. To identify biomarkers of response we will correlate ORR and PFS with ARID1A gene alteration, ARID1A protein level (IHC and DSP), gammaH2AX (IHC and DSP), C-myc (DSP), and total (tot) ATM (DSP), and HEXIM1 by ribonucleic acid (RNA) sequencing (Seq) in tumor biopsies (PART II).

X. To explore if liquid biopsies are a good surrogate for tumor ARID1A pathogenic alteration (PART II).

XI. To evaluate if ARID1A expression changes over time, we will compare ARID1A expression by NGS (gene alteration) and IHC (protein) using existing archival tumor to most recent pre-treatment biopsy samples required for PART II expansion cohort (PART II).

OUTLINE: This is a dose-escalation study of tuvusertib followed by a dose-expansion study.

Patients receive tuvusertib and BET bromodomain inhibitor ZEN-3694 orally (PO) on study. Patients in the dose-escalation phase of the trial also undergo electrocardiography (ECG) during screening, collection of blood samples on study, and x-ray, computed tomography (CT), or magnetic resonance imaging (MRI) throughout the trial. Patients in the dose-expansion phase of the trial also undergo ECG during screening, biopsies during screening and on study, and x-ray, CT, or MRI, and collection of blood samples throughout the trial.

After study completion, patients are followed every 3 months for 2 years and then every 6 months for 3 years, or until the study is terminated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pathologically confirmed:

  * PART I: Recurrent clear cell or endometrioid ovarian carcinoma (at least 50% morphology of clear cell and endometrioid required), recurrent clear cell and low grade endometrioid endometrial carcinoma (The International Federation of Gynecology and Obstetrics [FIGO] grade 1), or recurrent platinum resistant high grade serous ovarian carcinoma
  * NOTE: platinum-resistant disease is defined as progression within < 6 months from completion of platinum-based therapy. The date should be calculated from the last administered dose of platinum therapy
  * NOTE: Institutional pathology reports must be provided indicating at least 50% endometrioid or clear cell morphology for ovarian cancer.
  * NOTE: Patients with recurrent endometrial carcinoma must not be eligible for or decline treatment with curative intent.
  * PART II: Recurrent clear cell or endometrioid ovarian carcinoma (at least 50% tumor morphology of clear cell and endometrioid required). Recurrent clear cell or FIGO Grade 1 endometrioid endometrial carcinoma. Next Generation Sequencing (NGS) by Clinical Laboratory Improvement Act (CLIA) approved lab required for ARID1A status. Tumor will be determined as ARID1A pathologic alteration or likely pathologic alteration (Cohort I) or ARID1A wildtype by NGS (Cohort II). The number of patients in PART II cohort with clear cell or endometrioid EMCA will be capped at 33% (5 patients per cohort). Institutional pathology reports must be provided indicating at least 50% endometrioid or clear cell morphology for ovarian cancer.
* Age >= 18
* Eastern Cooperative Oncology Group (ECOG) Performance Status of =< 2
* Prior Treatment

  * 1-3 prior cytotoxic therapies

    * NOTE: For platinum-resistant HGSOC (PART 1) may have received up to 3 prior cytotoxic therapies after developing platinum resistant disease.
  * Subjects with microsatellite instability- high (MSI-H) and/or mismatch repair protein deficient (dMMR) endometrioid endometrial cancer must have previously received an immune checkpoint inhibitor.
  * Unlimited prior hormonal therapy, targeted therapy (including immunotherapy), and/or antiangiogenic therapy will be permitted.
* Washout periods (due to risk of myelosuppression):

  * Cytotoxic chemotherapy - 3 weeks.
  * Radiation therapy - 2 weeks (NOTE: patients with radiation to > 25% of the bone marrow are NOT eligible).
* Disease status:

  * For PART I, evaluable disease or measurable disease required. NOTE: evaluable disease: defined as disease related abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions.
  * For PART II, measurable disease by RECIST 1.1 is required. Patients will be required to undergo biopsy, which may be a non-target lesion but should not be the only RECIST measurable lesion.

NOTE: Patients for PART II are required to undergo paired tumor biopsies. If at time of biopsy the biopsy is deemed unsafe by interventional radiology or attempted and is unsuccessful, patients may still enroll.

* Hemoglobin >= 9 g/dL (in the absence of transfusion within 28 days prior to dosing)
* Absolute neutrophil count >= 1,500 cells/mm^3
* Platelet count >= 100,000 cells/mm^3
* Calculated creatinine clearance (CrCL) of >= 50 mL/min by the Cockcroft-Gault formula
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (patients with known Gilbert's disease who have bilirubin level =< 3 x ULN may be enrolled)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x institutional ULN
* Patients with known history or current symptoms of cardiac disease or history of treatment with cardiotoxic agents should be New York Heart Association (NYHA) Functional Classification of class I or II.
* The effects of M1774 and ZEN003694 on the developing human fetus are unknown. For this reason and because BETi agents are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately. Women of reproductive potential should use effective contraception treatment with M1774 and ZEN003694 and for at least 6 months following the last dose. Women should be advised not to breastfeed while taking M1774 and ZEN003694 and for 1 month after cessation of treatment.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with treated brain metastases are eligible if follow up brain imaging after central nervous system (CNS) directed therapy shows no evidence of progression, are off steroids, and are stable for at least 1 month.
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information.
* PART II only: Participants must have known mutational status (wild-type or pathogenic or likely pathogenic alteration) for ARID1A by Next-Generation Sequencing. This can be determined according to local testing generated by an assay with appropriate regulatory status.
* Patients must be able to swallow oral medications (capsules and tablets) without chewing, breaking, crushing, opening, or otherwise altering the product formulation.
* Patients with co-morbidities:

  * Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
  * For patients with evidence of chronic Hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
  * Patients with a history of Hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load.
* Resolution of all toxicities of prior therapy or surgical procedures to baseline or grade 1 (except for hypothyroidism requiring medication, which must have resolved to Grade =< 2), alopecia, and other toxicities considered clinically nonsignificant and/or stable on supportive therapy as determined by the investigator).

Exclusion Criteria:

* Patients who are receiving any other investigational agents.
* Patients who have received prior ATR, ATM, CHK, BET, EZH2, and/or PI3K inhibitors.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ZEN003694 or M1774 used in study.
* Patients taking proton pump inhibitors given decreased solubility of M1774 with increased pH. Proton pump inhibitors must be discontinued 7 days prior to initiating the trial.
* Patients with corrected QT (QTc) over 450msec that does not correct with correction of electrolyte abnormalities or family history of long QT syndrome.
* Patients with severe, active co-morbidity defined as follows:

  * No active infection requiring parenteral antibiotics.
  * Known hereditary diseases characterized by genetic defects of DNA repair mechanisms, including ataxia telangiectasia, Nijmegen breakage syndrome, Werner syndrome, Bloom Syndrome, Fanconi anemia, xeroderma pigmentosum, Cockayne syndrome, and trichothiodystrophy.
* Pregnant and breastfeeding women are excluded from this study because ZEN003694 has the potential for teratogenic or abortifacient effects and M1774 is genotoxic in in vivo nonclinical studies. Patients who discontinue breastfeeding are eligible for enrollment and may not resume breastfeeding until 1 month off treatment.
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible. Strong inhibitors or inducers of CYP3A4 must be discontinued at least 7 days prior to the first dose of ZEN003694. Moderate inhibitors of CYP3A4 should be avoided. If alternative is not available, the use of moderate CYP3A4 inhibitors is permitted with careful monitoring and approval by study team. At the discretion of the provider, additional monitoring (labs, toxicity checks) may be implemented for use of moderate CYP3A4 inhibitors. Substrates of CYP1A2 with narrow therapeutic window also must be avoided white taking ZEN003694. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product.
* Patients receiving any medications or substances that are Factor Xa inhibitors are discouraged given concerns for thrombocytopenia (i.e., rivaroxaban, apixaban, betrixaban, edoxaban otamixaban, letaxaban, eribaxaban) and Factor IIa inhibitors (i.e., dabigatran). Low molecular weight heparin is allowed. If patients are not willing to switch to low molecular heparin, they must obtain approval by study team.
* Serious gastrointestinal bleeding within 3 months, refractory nausea and vomiting, uncontrolled diarrhea, known malabsorption, significant small bowel resection or gastric bypass surgery, use of feeding tubes, presence of drainage gastrostomy tube, other chronic gastrointestinal disease, and/or other situations that may preclude absorption of oral medications M1774 and/or ZEN003694.
* M1774 restrictions:

  * Patients who cannot discontinue drugs that are strong inhibitors of CYP3A4 or CYP1A2.
  * Patients who cannot discontinue drugs that use hMATE1 or hMATE2-K substrates.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicities (DLTs) (Part I) | Within the first cycle of study treatment (up to 28 days)
  DLT is defined as any adverse events considered possibly, probably or definitely related to study drug combination as evaluated by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0. A Bayesian Optimal Interval (BOIN) design will be used to determine the MTD (Yuan et al. 2016). Will be summarized by dose level.
DLTs (Part II) | Within the first 2 cycles of study treatment (up to 56 days)
  DLT is defined as any adverse events considered possibly, probably or definitely related to study drug combination as evaluated by NCI CTCAE v5.0. Within the ARID1A cohorts, the number of patients with DLTs will be summarized, and adverse events tabulated using the highest observed grade for each system organ class or preferred term, using CTCAE v5.0 criteria by cohort.
Measurements for gammaH2AX (PART II) | Baseline and cycle 1, day 8 (C1D8)
  GammaH2AX will be assessed by immunohistochemistry (IHC) from tumor samples. Will be summarized using descriptive statistics (e.g., mean, standard deviation, median) by cohort and collection time point. One-sided Wilcoxon signed rank tests will be used for testing whether there is a change in gammaH2AX expression in the pre-treatment vs on-treatment tumor in the patients who have been treated at the recommended phase 2 dose (RP2D) and have evaluable bio-specimen by cohort, respectively.
Incidence of adverse events (Part I and II) | Up to 5 years
  The frequency and severity of adverse events will be assessed by CTCAE v5.

SECONDARY OUTCOMES:
Measurements for c-myc (Part II) | Baseline and C1D8
  Will be assessed by Digital Spatial Profiling (DSP) using tumor samples. Will be summarized using descriptive statistics (e.g., mean, standard deviation, median) by cohort, biospecimen type, and collection time point. One-sided Wilcoxon signed rank tests will be applied to examine whether there is a change in c-myc expression in the pre-treatment vs on-treatment tumor in the patients who have been treated at the RP2D and have evaluable bio-specimen by cohort, respectively.
Measurements for gammaH2AX (Part II) | Baseline and C1D8
  Will be assessed by DSP using tumor samples. Analyses will be performed in similar approach to the primary endpoint gammaH2AX expression by IHC.
Measurements for ARID1A protein and pathogenic alteration status (Part II) | Baseline, C1D8, and at progression
  Summary statistics (e.g., mean and standard deviation, median) for ARID1A protein by IHC and DSP in pre-treatment tumor will be provided for the 12-point score (measure of ARID1A positive staining cells by IHC) by cohort and mutation status (Khalique et al, 2018). ARID1A pathogenic alteration means there is loss of ARID1A protein as assessed by IHC and DSP. ARID1A wildtype means there is no mutation and ARID1A protein is present. The relationship between ARID1A protein and ARID1A pathogenic alteration status will be investigated by Wilcoxon rank-sum test.
Objective response rate (Part II) | At 6 months
  Objective response rate (ORR) is defined as the binomial proportion of evaluable patients with best overall response assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 of complete or partial response (CR or PR).
Progression-free survival (Part II) | From study entry to time of progression or death, whichever occurs first, or date of last contact if neither progression nor death has occurred, assessed at 6 months
  Progression-free survival at six months (PFS) is defined as the binomial proportion of evaluable patients who survive without documentation of disease progression (RECIST 1.1) at least 6 months after starting study entry.

OTHER OUTCOMES:
Measurements of blood pharmacokinetics (PK) for ZEN003694 and ZEN003791 (Part I) | C1D1 (Pre-dose, 0.5, 1, 1.5, 2, 3, 4, & 8 hours [hrs]); C1D8 (Pre-dose, 0.5, 1, 1.5, 2, 3, 4, & 8 hrs)
  PK endpoints (area under the curve [AUC], maximum concentration [Cmax] and metabolic ratio of ZEN003694 and active metabolite ZEN003791, and M1774) will be summarized using descriptive statistics by dose level.
Measurements for ARID1A protein (Part I) | Baseline
  ARID1A status and molecular profiles will be tabulated retrospectively.
Objective response rate (Part I) | At 6 months
Progression-free survival (Part I) | From study entry to time of progression or death, whichever occurs first, or date of last contact if neither progression nor death has occurred, assessed at 6 months
Measurements of biomarker molecular profile (Part I) | Up to 5 years
  Will assess profiles by Next Generation Sequencing from somatic tumor, correlate other molecular alterations (e.g., PIK3CA, C-Myc) with response by RECIST 1.1 and CA-125 by Gynecological Cancer Intergroup (GCIG).
Measurements of blood PK for ZEN003694 and ZEN003791 when taken alone or with M1774 (Part II) | C1D1 (Pre-dose & 2 hrs); C1D8 (2 hrs)
  Will be summarized using descriptive statistics by dose level and non-linear model techniques.
Correlation of objective response rate, CA-125 response, and overall survival (OS) with ARID1A pathogenic alteration status (Part II) | Up to 5 years
  Objective tumor response (complete or partial response) by RECIST 1.1 and GCIG CA-125 will be tabulated by cohort, respectively, and the proportion of patients with response will be estimated and compared between the two cohorts by Fisher's exact test.
Correlation of measurements for PK and pharmacodynamics (e.g., gH2AX and MYC) (Part II) | Up to 5 years
  Descriptive statistics or mixed modeling approaches may be used to explore the corresponding associations of pharmacodynamic biomarkers with PK plasma concentration for ZEN003694.
Measurements for ARID1A genetic status, ARID1A protein level, gammaH2AX, c-myc, total ATM, HEXIM1 | Up to 5 years
  Will assess ARID1A protein level (IHC and DSP), gammaH2AX (IHC and DSP), c-myc (DSP), total ATM (DSP), HEXIM1 by ribonucleic acid sequencing (RNASeq) in tumor biopsies, and correlation with objective response rate, and progression-free survival. Will be explored by Spearman's correlation coefficient, respectively.
Correlation of ARID1A gene alteration in circulating free tumor deoxyribonucleic acid (ctDNA) with tumor ARID1A genetic status and protein expression | Up to 5 years
  Summary statistics for ARID1A genetic status from pre-treatment blood specimen will be provided, and the associations of it with tumor ARID1A genetic status and protein expression from pre-treatment biopsies, and objective tumor response will be explored by appropriate non-parametric methods, e.g., Spearman's correlation coefficient methods for ordinal-type data.
Measurements for ARID1A expression | At pre-treatment
  Will be assessed by NGS (gene alteration) and IHC from archival tumor and compare to most recent pre-treatment biopsy. The ARID1A genetic status and protein in archival tumor and most recent pre-treatment biopsy will be summarized by time, and the corresponding changes will be explored using Wilcoxon's signed rank tests or repeated measures methods.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Simpkins, Principal Investigator — NRG Oncology
Locations (14):
- United States (14):
  - Augusta University Medical Center, Augusta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - NRG Oncology, Philadelphia, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm